CLINICAL TRIAL: NCT00242983
Title: Assessment of Quality of Life (QOL) in Patients Registered With "Phase III Randomized Comparison Study of Vinorelbine, Gemcitabine, and Docetaxel Versus Paclitaxel and Carboplatin in Patients With Advanced Non-Small Cell Lung Cancer (JMTO LC00-03)"
Brief Title: Quality of Life in Patients Who Are Receiving Either Vinorelbine, Gemcitabine, and Docetaxel or Paclitaxel and Carboplatin for Advanced Non-Small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Hospital Organization Kinki-chuo Chest Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000450163; NHOK-BRI-LC03-01
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2005-12

CONDITIONS: Lung Cancer
Keywords: adenocarcinoma of the lung; large cell lung cancer; recurrent non-small cell lung cancer; squamous cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung

INTERVENTIONS:
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Studying quality-of-life in patients undergoing cancer treatment may help identify the intermediate and long-term effects of treatment on patients with cancer.

PURPOSE: This clinical trial is studying quality of life in patients who are receiving either vinorelbine, gemcitabine, and docetaxel or paclitaxel and carboplatin for advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the quality of life of patients with advanced non-small cell lung cancer treated with vinorelbine, gemcitabine, and docetaxel vs paclitaxel and carboplatin on protocol JMTO-LC00-03.

OUTLINE: This is a multicenter study. Patients receive treatment on protocol JMTO-LC00-03.

Quality of life is assessed using the Functional Assessment of Cancer Therapy-Lung (FACT-L), FACT-Taxane, and Functional Assessment of Chronic Illness Therapy-Spirituality (FACIT-Sp) questionnaires at baseline, weeks 9 and 18, and at the completion of treatment.

PROJECTED ACCRUAL: A total of 80 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed primary non-small cell lung cancer, including any of the following:

  * Newly diagnosed selected stage IIIB (T4 lesion due to malignant pleural effusion) disease
  * Newly diagnosed stage IV disease
  * Recurrent disease after prior surgery and/or radiotherapy
* Any of the following cellular subtypes are allowed:

  * Adenocarcinoma
  * Large cell carcinoma
  * Squamous cell carcinoma
  * Unspecified carcinoma
* Enrolled on protocol JMTO-LC00-03

PATIENT CHARACTERISTICS:

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY:

Radiotherapy

* See Disease Characteristics

Surgery

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-04

PRIMARY OUTCOMES:
Change in the total score from baseline measured by the Functional Assessment of Cancer Therapy-Lung (FACT-L), FACT-Taxane, and Functional Assessment of Chronic Illness Therapy-Spirituality (FACIT-Sp) questionnaires at 9, 18, and 22 weeks or withdrawal

SECONDARY OUTCOMES:
Change in the subscale from baseline of these questionnaires at 9, 18, and 22 weeks or withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Masaaki Kawahara, MD, Study Chair — National Hospital Organization Osaka National Hospital
Locations (21):
- Japan (21):
  - Toyohashi Municipal Hospital, Aichi
  - Ichinomiyanishi Hospital, Aichi
  - Asahikawa Medical College, Asahikawa
  - National Cancer Center Hospital East, Chiba-ken
  - Shikoku Cancer Center Hospital, Ehime
  - National Hospital Organization - Nishigunma National Hospital, Gumna
  - Gunma Cancer Center, Gunma
  - National Hospital Organization - Dohoku National Hospital, Hokkaido
  - Junshinkai Tsuna Hospital, Hyōgo
  - Takarazuka Municipal Hospital, Hyōgo
  - Fujisawa City Hospital, Kanagawa
  - National Hospital Organization - Minamikyoto Medical Center, Kyoto
  - Miyagi Cancer Center, Miyagi
  - National Hospital Organization - Okayama Medical Center, Okayama
  - Osaka Kosei Nenkin Hospital, Osaka
  - Osaka General Medical Center, Osaka
  - National Hospital Organization - Osaka National Hospital, Osaka
  - Saitama Cardiovascular and Respiratory Center, Saitama
  - Tokyo Medical University, Tokyo
  - Tottori University Hospital, Tottori
  - Koseiren Takaoka Hospital, Toyama

REFERENCES:
- [Derived] Kawahara M, Tada H, Tokoro A, Teramukai S, Origasa H, Kubota K, Shinkai T, Fukushima M, Furuse K. Quality-of-life evaluation for advanced non-small-cell lung cancer: a comparison between vinorelbine plus gemcitabine followed by docetaxel versus paclitaxel plus carboplatin regimens in a randomized trial: Japan Multinational Trial Organization LC00-03 (BRI LC03-01). BMC Cancer. 2011 Aug 17;11:356. doi: 10.1186/1471-2407-11-356. PMID 21849041